CLINICAL TRIAL: NCT03411239
Title: Assessment of Airway Pressure Changes Using Esophageal Balloon Catheter (OBC) in Patients Undergoing Laparoscopic Surgery Under General Anaesthesia
Brief Title: Airway Pressure Changes Using Esophageal Balloon Catheter (OBC) in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/00153
Record Dates: First submitted 2017-09-19; First posted 2018-01-26 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2021-10

CONDITIONS: Ventilator Lung
Keywords: Airway pressure; Oesophageal pressure; transpulmonary pressure; laparoscopic surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Other): Patients recruited will have OBC inserted under general anaesthesia and various pressure measured
  Interventions: Device: Adult esophageal balloon catheter (obc)

INTERVENTIONS:
Device: Adult esophageal balloon catheter (obc) — Using OBC to determine airway pressure changes in patients undergoing general anaesthesia for laparoscopic surgery

SUMMARY:
This is a single centre study. The investigators intend to recruit 20 subjects over 4 months. Patients undergoing laparoscopic abdominal surgery for cholecystectomy, laparoscopic gynaecological surgery and laparoscopic urologic procedures either as day surgery, same day admission or in patients, will be included in the study. Patients will be identified at the time of listing for surgery and referred to study team, which in turn will recruit the patients. Informed consent will be obtained at the time of recruitment and a copy of consent with details of principal investigator would be provided to subjects. All data collection will be done intraoperative. Patient would be followed up once at day 3 post op period. If patients have any complications related to the study, they will be followed up weekly until the complication is resolved.

DETAILED DESCRIPTION:
General anaesthesia: Patients will be induced and intubated as per the choice of consultant anaesthetist. Anaesthesia will be maintained with inhalational agent and paralysis maintained with atracurium infusion or bolus so as to keep train of four counts <2 twitches using peripheral nerve stimulator throughout surgery. Conventional ventilation was standardised with mode as pressure control ventilation, pressure inspired targeted to either tidal ventilation of 6-8 ml/kg or end tidal carbon di oxide concentration of 40-50 mmHg and positive end expiratory pressure limited to 5 cm of water. Fraction of inspiratory oxygen was adjusted to keep oxygen saturation > 95%. No recruitment manoeuvres were permitted unless, patient is desaturating actively, and in which case patient will be excluded from the study. Abdominal cavity was insufflated with carbon dioxide with initial high flow and pressure, but later the pressure was maintained at 15cm water.

Esophageal balloon catheter insertion, placement and removal: After applying topical anaesthetic (10% lidocaine spray) to patient's nasopharynx and water-soluble lubricant jelly to distal end of esophageal catheter, it is inserted into patient's esophagus via nasal cavity or oropharyngeal cavity. Estimated depth of catheter insertion is calculated as: patient's height (in cm) X 0.288. Once the esophageal balloon catheter is inserted to estimated depth, balloon is inflated with 4 ml of air and pressure on the stomach is applied to look for positive deflection of oesophageal pressure reading. Once convinced, 2 ml air was taken out and catheter was slowly withdrawn till cardiac oscillations are visible. Occlusion test is performed to confirm the placement of catheter in lower thoracic region. In occlusion test, patient is briefly disconnected from ventilator, endotracheal tube is blocked and pressure is applied on to chest wall. Simultaneous increase in oesophageal balloon pressure and airway pressure is noted. (Change is oesophageal pressure/ change in airway pressure on application of external pressure should be close to 1). Stylet is removed and Oesophageal balloon catheter is secured at this position on nostril or angle of mouth similar to nasogastric tube and connected to pressure transducer to do necessary measurements. Catheter is removed at the end of surgery before extubation after complete deflation of cuff.

Measurements: Soon after confirmation of position, patient is subjected to end inspiratory hold to record the end inspiratory pleural pressure and plateau airway pressure. Patient is then subjected to end expiratory hold to record end expiratory pleural pressure and positive end expiratory pressure. Similar steps are repeated once pneumoperitoneum is achieved and patient is placed in trendelenburg or reverse trendelenburg position and once pneumoperitoneum deflated. Problems encountered during insertion and measurement of esophageal balloon catheter will be resolved using manufacturer's recommendation.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade 1 and 2 patients,
2. Age > 21 yrs.
3. Elective intraabdominal laparoscopic surgery

Exclusion Criteria:

1. ASA grade 3 and 4 patients
2. Emergency surgery
3. Patient with tracheostomy
4. Patient with any oropharyngeal pathology
5. Patients with co-existing respiratory disease i.e. COPD, restrictive lung disease.
6. Patients with oesophageal diseases: varicose, stricture, recent esophageal or gastric surgery.
7. Patients with nasopharyngeal diseases: sinusitis, epistaxis, nasopharyngeal carcinoma post radiotherapy or chemotherapy.
8. Age < 21 years
9. Pregnant females

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Inspiratory and expiratory oesophageal pressure during laparoscopic surgery | 1 year
  using pressure monitoring line
Inspiratory and expiratory transpulmonary pressure during laparoscopic surgery | 1 year
  difference between oesophageal pressure and airway pressures
Inspiratory and expiratory transpulmonary pressure during supine, trendelenburg and reverse trendelenburg position | 1 year
  difference between esophageal pressure and airway pressure in various positions

CONTACTS AND LOCATIONS:
Overall Officials: Rohit V Agrawal, MMed, FANZCA, Principal Investigator — Consultant, Department of Anaesthesia, NUH
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, results, analysis